CLINICAL TRIAL: NCT07005245
Title: The Demand for Psychological and Social Services Related to COVID-19 Pandemic in Families of Patients With Severe Mental Disorders
Brief Title: Survey on the Reproductive and Child-Rearing Situations of Patients With Severe Mental Disorders
Status: Completed | Type: Observational
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-1-13-7
Record Dates: First submitted 2025-05-19; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2021-01

CONDITIONS: Schizophrenia and Schizoaffective Disorder; Bipolar Disorder (BD)
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional

SUMMARY:
Severe mental disorders represent a major public health concern, imposing substantial disease burden and adversely affecting multiple dimensions of patients' lives, while also creating intergenerational impacts on their offspring and families. Existing evidence suggests that children of affected patients demonstrate elevated vulnerability to various physical and psychological challenges during developmental stages.

Currently, China lacks systematic data regarding reproductive patterns and child-rearing practices among patients with severe mental disorders. To address this knowledge gap, investigators are conducting a multicenter epidemiological survey across ten representative cities and regions nationwide. This study aims to comprehensively examine the reproductive history, child-rearing circumstances, and family socioeconomic status of this population. The findings will establish a crucial foundation for subsequent analytical epidemiological investigations and intervention studies, while informing evidence-based mental health policy formulation.

The study population consists of registered patients (aged 18-59 years) in the national severe mental disorder management system who meet diagnostic criteria for: schizophrenia, bipolar disorder, paranoid personality disorder, schizoaffective disorder, epilepsy-induced mental disorders, or intellectual disability-associated mental disorders. Eligible participants must have documented childbirth history (including miscarriage, preterm, and term deliveries).

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the diagnostic criteria for schizophrenia, bipolar disorder, paranoid personality disorder, schizoaffective disorder, mental disorders caused by epilepsy, or mental disorders associated with intellectual disabilities, and are registered in the management system for severe mental disorders
* Aged 18-60 years
* Patients who had a history of childbirth (childbirth history includes miscarriage, preterm birth, and full-term birth).

Exclusion Criteria:

* Do not agree to participate in the survey.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Peking University Sixth Hospital, 51 Huayuan North Road, Haidian District, Beijing.
Sampling Method: Non-Probability Sample
Enrollment: 77145 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Participants' fertility data | Baseline

SECONDARY OUTCOMES:
Somatic/psychiatric morbidity history in participants' offspring | Baseline

OTHER OUTCOMES:
Participants' demographics, their offspring's education level, and family caregiving situation | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Sixth Hospital, Beijing, Haidian District, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sheng Z, Zhou T, Du C, Wu T, Wen L, Yang X, Chen W, Ma X, Deng H, Ge L, Zhang C, Hong X, He R, Du X, Zhu L, Xiang H, Chen S, Liu J, Ding Y, Liang G, Pan Y, Ji S, Chang Z, Yuan N, Chen W, Lv X, Ma H, Guan L, Yu X. Sex-differences in the intergenerational transmission of mental disorders among schizophrenia probands: familial risk and protective factors in a population-based study. Lancet Reg Health West Pac. 2025 Nov 20;65:101750. doi: 10.1016/j.lanwpc.2025.101750. eCollection 2025 Dec. PMID 41362421

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/45/NCT07005245/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/45/NCT07005245/ICF_001.pdf